CLINICAL TRIAL: NCT00505999
Title: Etiology of Multiple Myeloma: A Case-Control Study
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2006-0141; R25CA057730 (NIH)
Record Dates: First submitted 2007-07-24; First posted 2007-07-25 (Estimated); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Etiology; Risk Factors; Healthy Controls; Questionnaire; Survey
MeSH Terms: conditions — Multiple Myeloma | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and saliva samples that will be used for special tests to look for any biological factors associated with Multiple Myeloma (MM).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

GROUPS / COHORTS (1):
- Questionnaire: Patients diagnosed with Multiple Myeloma and healthy controls.
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — Questionnaire taking 30-40 minutes to complete.
  Other Names: Survey

SUMMARY:
Objectives:

The overall objective of this project is to identify risk factors associated with the development of multiple myeloma (MM) by integrating epidemiologic, clinical and molecular information. We plan to invite MDACC patients with MM, as well as controls, to participate in this investigative case-control study. Controls will be selected from friends and spouses who accompany patients to the various MDACC clinics and will be matched to the cases on age (±5 years), gender, and ethnicity. We will obtain demographic, risk factor and clinical information along with a blood and buccal sample from all cases and controls. This study could have implications for prevention and subsequent reduction in the incidence of multiple myeloma. Collecting blood and buccal samples will allow us to study the role genetic susceptibility plays in MM risk. The specific aims are:

1. To enroll and obtain, through self-administered questionnaires, risk factor information on all study participants to develop detailed demographic, epidemiologic, and behavioral profiles. This study will accrue 250 MM patients from MDACC and 250 healthy controls selected from friends and spouses who accompany patients to the MDACC clinics. Blood (25 ml) and buccal samples will be collected from all participants.
2. To identify risk factors associated with MM by integrating epidemiological, clinical and molecular information using a case-control approach.
3. To evaluate constitutional markers of genetic susceptibility as predictors of MM risk. Gene-environment interactions will be explored.

DETAILED DESCRIPTION:
Informed Consent For Control Subjects:

In this study, researchers are trying to learn about factors that may be associated with MM.

For this study, you will be asked to complete a questionnaire. The questionnaire asks questions about your demographics (for example, age and sex), any chemicals you may have been exposed to, your medical history, family history of cancer, your diet, and your history of smoking and/or alcohol use. It should take around 30-40 minutes to complete the questionnaire.

Blood (about 2-3 tablespoons) will be drawn. You will spit into a collection container in order to provide a sample of your saliva. The blood and saliva samples will be used for special tests to look for any biological factors associated with MM.

If you live in Houston or the surrounding area, study personnel can arrange to collect the samples at the time and place of your convenience. If you do not live in the Houston area, sample collection instructions and supplies will be mailed to you. The blood sample may be drawn at your doctor's office, or at a clinic or hospital of your choice. All mailing costs will be paid by the study. No travel to M. D. Anderson will be required.

You will be considered off-study after the data that is collected has been processed.

This is an investigational study. Up to 500 participants will take part in this study. All will be enrolled at M. D. Anderson.

Informed Consent for Patients:

In this study, researchers are trying to learn about factors that may be associated with MM.

For this study, you will be asked to complete a questionnaire. The questionnaire asks questions about your demographics (for example, age and sex), any chemicals you may have been exposed to, your medical history, family history of cancer, your diet, and your history of smoking and/or alcohol use. It should take around 30-40 minutes to complete the questionnaire.

Blood (about 2-3 tablespoons) will be drawn. You will spit into a collection container in order to provide a sample of your saliva. The blood and saliva samples will be used for special tests to look for any biological factors associated with MM.

If you live in Houston or the surrounding area, study personnel can arrange to collect the samples at the time and place of your convenience. If you do not live in the Houston area, sample collection instructions and supplies will be mailed to you. The blood sample may be drawn at your doctor's office, or at a clinic or hospital of your choice. All mailing costs will be paid by the study. No travel to M. D. Anderson will be required.

Neither you nor your doctor will receive the results of these tests, and they will not be put in your medical record.

You will be considered off study after the data that is collected has been processed.

This is an investigational study. Up to 500 participants will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Cases: MDACC patients with confirmed MM who consent to complete a risk factor questionnaire and donate a 25ml blood specimen and a buccal sample.
2. Controls: Friends or spouses of MDACC patients matched on age (± 5 years), sex and ethnicity who consent to complete a risk factor questionnaire and donate a 25 ml blood specimen and a buccal sample.

Exclusion Criteria:

1. Cases: No exclusion criteria.
2. Controls: Previous history of invasive cancer (excluding non-melanoma skin cancer)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with Multiple Myeloma and healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2006-07 (Actual); Primary Completion 2020-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
The goal of this epidemiological research study is to identify biological and lifestyle factors that may be associated with the development of Multiple Myeloma (MM). | 2 Years

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Hildebrandt, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: The University of Texas M.D.Anderson Cancer Center — http://www.mdanderson.org